CLINICAL TRIAL: NCT00287664
Title: Terlipressin as Treatment of Patients With Cirrhosis and Hepatorenal Syndrome. Effect on Survival and Renal Function. Multicenter, Randomized and Prospective Study
Brief Title: Treatment of Hepatorenal Syndrome With Terlipressin Plus Albumin vs Albumin
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: because in a preliminary analysis we would need 1000 patients per group to achieve significative differences in the main end point.
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Grant from Education Ministery from 2001-2004. (Unknown)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TAHRS
Record Dates: First submitted 2006-02-03; First posted 2006-02-07 (Estimated); Last update posted 2007-04-11 (Estimated); Status verified 2007-04

CONDITIONS: Cirrhosis; Hepatorenal Syndrome
Keywords: hepatorenal syndrome; terlipressin; albumin; cirrhosis
MeSH Terms: conditions — Fibrosis; Hepatorenal Syndrome | interventions — Terlipressin

INTERVENTIONS:
Drug: terlipressin

SUMMARY:
Hepatorenal syndrome is a common complication of cirrhotic patients. The prognosis of patients with HRS is very poor. It have been demonstrated that vasoconstrictors agents (Terlipressin) plus albumin are effective in the reversal of the treatment. However, previous studies are pilot studies and they are not able to give information about an improvement in survival. This comparative randomized study was delineated to test the efficacy of terlipressin on survival.

DETAILED DESCRIPTION:
Phase 3

ELIGIBILITY:
Inclusion Criteria:

1. Patients with HRS type 1 or 2 with serum creatinine >2 mg/dL
2. Age between 18 and 75 years
3. Written informed consent.
4. Absence of exclusion criteria

Exclusion Criteria:

1. Hepatocarcinoma (3 nodules greater than 3 cm or 1 nodule > than 5 cm)
2. Active infection with systemic inflammatory response syndrome
3. Respiratory or cardiac dysfunction.
4. Arteriopathy.
5. Ischemic cardiopathy.
6. Arterial hypertension ( >140/90 mmHg during hospitalization )

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2002-02; Study Completion 2006-09

PRIMARY OUTCOMES:
Survival

CONTACTS AND LOCATIONS:
Overall Officials: Pere Gines, MD, Principal Investigator — Chair of Liver Unit
Locations (1):
- Hospital Clinic, Barcelona, Barcelona, Spain